CLINICAL TRIAL: NCT01368744
Title: Intraoperative Examination of Sentinel Lymph Nodes: Comparison of the OSNA Breast Cancer System to Extensive Frozen Section Histopathology
Brief Title: Clinical Evaluation of OSNA Breast Cancer System to Extensive Frozen Section Histopathology
Status: Completed | Type: Observational
Sponsor: Sysmex America, Inc. (Industry)
Responsible Party: Carrie Pineda, Sysmex America, Inc
Other Study IDs: OSNA-BC-002
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Breast Neoplasms; Breast Diseases
Keywords: Breast Neoplasms; Breast Diseases
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of the tissue homogenate will be retained and may be used for for further testing.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- OSNA Breast Cancer System
  Interventions: Device: OSNA Breast Cancer System

INTERVENTIONS:
Device: OSNA Breast Cancer System — For in vitro diagnostic use only.
  The OSNA Breast Cancer System is an automated semi-quantitative, in vitro diagnostic test for the rapid detection of greater than (>) 0.2 mm metastases in nodal tissue removed from sentinel lymph node biopsies of breast cancer patients. Results from the assay can be used to guide the intra-operative or post-operative decision to remove additional lymph nodes and to aid in patient staging. An assay positive + or ++ result indicates the presence of metastasis (> 0.2 mm). An assay positive ++ result predicts the presence of macrometastasis (> 2 mm).
  Groups: OSNA Breast Cancer System

SUMMARY:
The study will determine the sensitivity, specificity, negative predictive value and positive predictive value of the OSNA Breast Cancer System by comparing its performance to an extensive intraoperative frozen section protocol for Sentinel Lymph Nodes removed during standard Sentinel Lymph Node biopsy procedures from breast cancer subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* 18 years of age or older;
* Diagnosed pre-surgically with T1 or T2 breast cancer without clinical evidence of axillary lymph node involvement and scheduled for surgery including sentinel lymph node dissection;
* Subjects (or the subjects' legal representatives) who have read, understood to the best of their ability and signed the informed consent form.

Exclusion Criteria:

* Subjects diagnosed pre-surgically with large or locally advanced (T3 & T4) breast cancer;
* Pregnant subjects, confirmed by interview with either subject or treating physician;
* Subjects diagnosed with inflammatory breast cancer;
* Subjects diagnosed with ductal carcinoma in situ (DCIS) when breast conservation is to be done;
* Subjects with clinically suspicious, palpable axillary lymph nodes;
* Subjects previously treated for or previously diagnosed with another type of invasive cancer. Subjects with skin cancer (basal cell and squamous cell carcinoma) may be included, except for subjects diagnosed with melanoma; Subjects with non-invasive carcinoma of the Cervix may also be included in this study.
* Subjects who have received pre-operative systemic therapy;
* Subjects who are incapable of providing written informed consent;
* Subjects who have been judged to be an inappropriate candidate by any medical care provider (e.g., surgeon, oncologist or pathologist).
* Subjects participating in other clinical studies where the SLN evaluation will be negatively impacted by this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a previous diagnosis of breast cancer scheduled for sentinel lymph node dissection.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Prospectively assess the concordance and performance of the OSNA Breast Cancer System with an extensive intraoperative frozen section protocol for SLNs removed using standard SLN biopsy procedures from breast cancer subjects. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Milan School of Medicine, Milan, Italy, Italy